CLINICAL TRIAL: NCT04496336
Title: Non-invasive Substrate Evaluation in Atrial Fibrillation Using Cardiac Magnetic Resonance and Electrocardiographic Imaging
Brief Title: Non-invasive Substrate Evaluation in Atrial Fibrillation
Acronym: NOISE-AF
Status: Completed | Type: Observational
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Gregorio Marañón Hospital (Other)
Responsible Party: Principal Investigator, Josep Lluis Mont Girbau, Head of Arrythmia Unit, Hospital Clinic of Barcelona
Other Study IDs: NOISE-AF
Record Dates: First submitted 2020-07-29; First posted 2020-08-03 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: C14.280.067.198
Keywords: Atrial Fibrillation; Paroxysmal Atrial Fibrillation; Persistent Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims to assess the right and left atrial electrophysiological substrate in atrial fibrillation patients using the invasive electroanatomic map (basal and with extraestimulus) as well as its correlation with cardiac magnetic resonance and electrocardiographic imaging. The results will also be compared when the patient is in sinus rhythm and atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* Atrial fibrillation paroxysmal or persistent with criteria for percutaneous ablation

Exclusion Criteria:

* Cardiomiopathy (FEVI<40%) or significant valvulopathy.
* MRI not possible or contraindicated.
* Previous atrial fibrillation ablation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with persistent or paroxysmal atrial fibrillation, without cardiomyopathy (LVEF> 40%) or significant valvulopathy who will undergo first AF ablation.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2020-02-20 (Actual); Primary Completion 2022-10-20 (Actual); Study Completion 2022-11-20 (Actual)

PRIMARY OUTCOMES:
Correlation between conduction velocity and MRI fibrosis. | Baseline
  The conduction velocity in sinusal rhythm and with extra estimuli will be correlated with the MRI late gadolinium enhancement sequence (MRI-LGE).

SECONDARY OUTCOMES:
Correlation between voltage and MRI fibrosis. | Baseline
  The voltage in sinus rhythm and in atrial fibrillation will be correlated with the MRI-LGE.
Correlation between electrocardiographic image (ECGi) and MRI-LGE. | Baseline
  The xxx of the ECGi will be correlated with the MRI-LGE.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospital Gregorio Marañon, Madrid, Barcelona
  - Hospital Clinic de Barcelona, Barcelona